CLINICAL TRIAL: NCT01611883
Title: Examination of the Effect of Ezetimibe on Glucose Metabolism - Randomized, Double-blind, Placebo-controlled Study in Type 2 Diabetes Mellitus Patients With Hypercholesterolemia - Phase 4, Protocol No. 367 (Also Known as SCH 58235, P06541)
Brief Title: A Study of the Effect of Ezetimibe on Glucose Metabolism in Type 2 Diabetics With Hypercholesterolemia (P06541)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P06541; MK-0653-367 (Other: Merck Study Number)
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe (Experimental): 10 mg oral dose once daily for 24 weeks
  Interventions: Drug: Ezetimibe
- Placebo (Placebo Comparator): Placebo to match ezetimibe orally once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ezetimibe — 10 mg oral dose once daily for 24 weeks
  Other Names: MK-0653; SCH 058235
  Arms: Ezetimibe
Drug: Placebo — Placebo to match ezetimibe orally once daily for 24 weeks.
  Arms: Placebo

SUMMARY:
This study will examine the effect of ezetimibe on glucose metabolism in participants with Type 2 diabetes and hypercholesterolemia.The primary hypothesis is that change in glycated hemoglobin (HbA1c) from baseline in the ezetimibe treatment group will be non-inferior to the placebo control group.

ELIGIBILITY:
Inclusion Criteria:

* Have hypercholesterolemia (high cholesterol) and have been diagnosed with type 2 diabetes that is being treated with oral anti-diabetic drugs or insulin or both.
* No change in the medication (drugs, dose and administration) for the treatment of diabetes within previous 12 weeks with exception of small changes in insulin dosing
* No change in diet and exercise therapy within previous 4 weeks

Exclusion Criteria:

* Coexisting disease (hemoglobinopathy, hemolytic anemia, etc.) that may affect HbA1c measurement
* Homozygous or heterozygous familial hypercholesterolemia
* Previously received ezetimibe
* Hypercholesterolemia associated with: hypothyroidism, obstructive gall bladder or biliary disease, chronic renal failure or pancreatitis
* Hyperlipidemia caused by medication

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2014-01-16 (Actual); Study Completion 2014-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saito I, Azuma K, Kakikawa T, Oshima N, Hanson ME, Tershakovec AM. A randomized, double-blind, placebo-controlled study of the effect of ezetimibe on glucose metabolism in subjects with type 2 diabetes mellitus and hypercholesterolemia. Lipids Health Dis. 2015 May 1;14:40. doi: 10.1186/s12944-015-0036-z. PMID 25929253

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ezetimibe | Placebo
Started | 75 | 77
Completed | 74 | 76
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe | Placebo | Total
Number analyzed (Participants) | 75 | 77 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.8) | 60.0 (9.7) | 59.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 46 | 48 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Hemoglobin (HbA1c) From Baseline
Description: HbA1c is blood marker used to report average blood glucose levels over a prolonged period of time and is reported as a percentage (%). HbA1C was measured at baseline and after 24 weeks of study drug administration.
Time Frame: Baseline and Week 24
Population: Per Protocol Set defined as all randomized participants meeting inclusion criteria who were not excluded from the Full Analysis Set and were at least 75% compliant with study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 69 | 75
Percent | 0.22 [0.11 to 0.34] | 0.14 [0.03 to 0.25]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Non-Inferiority or Equivalence — Ezetimibe treatment group will be considered non-inferior to the placebo control group if the upper bound of the two-sided 95% confidence interval (CI) of the between-treatment difference (ezetimibe minus placebo) in means for change in HbA1c from baseline to the end of treatment does not exceed 0.5%; Longitudinal analysis of covariance; Treatment group, HbA1c level, insulin use, time, and "time × treatment group" interaction as factors, and baseline as covariate; Difference in Least-squares Means = 0.08, 95% CI 2-sided [-0.07 to 0.23] — ezetimibe minus placebo

2. Secondary Outcome: Change in Glycoalbumin From Baseline
Description: Glycoalbumin is a blood marker used to assess blood glucose control over time and is reported as a percentage (%). Serum glycoalbumin levels were assessed at baseline and after 24 weeks of study drug administration.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 69 | 75
Percent | -0.02 [-0.37 to 0.34] | -0.02 [-0.37 to 0.33]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; Longitudinal analysis of covariance; Difference in Least-squares Means = 0.00, 95% CI 2-sided [-0.47 to 0.47] — ezetimibe minus placebo

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline
Description: Plasma glucose levels were assessed after an overnight fast at baseline and after 24 weeks of study drug administration.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 69 | 75
mg/dL | 6.6 [1.1 to 12.1] | 11.4 [6.1 to 16.7]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; Longitudinal Analysis of Covariance; Difference in Least-squares Means = -4.8, 95% CI 2-sided [-12.1 to 2.5] — ezetimibe minus placebo

4. Secondary Outcome: Percentage of Participants With Adverse Event (AE) "Exacerbation of Diabetes"
Description: The Investigator took into account a participant's index of blood glucose control, diabetes medications, and compliance to diet and exercise therapy to assess overall control of the participant's diabetes and to determine if the participant's diabetes worsened. Participants who experienced the AE "Exacerbation of Diabetes " (verbatim term) were recorded.
Time Frame: up to 24 weeks
Population: All Subjects Treated (AST) Population defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 75 | 77
Percentage of Participants | 9.3 | 7.8
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Comparison of percentage difference between ezetimibe and placebo; Test type: Superiority or Other; p = 0.779, Fisher Exact

5. Secondary Outcome: Percentage of Participants With Changes in Diabetes Medications Due to Worsening of Diabetes
Description: The percentage of participants who had changes to their medications used to treat their diabetes, other than small changes in insulin dosing (± 5 Units), were reported and summarized.
Time Frame: Up to 24 weeks
Population: AST Population defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 75 | 77
Percentage of Participants | 9.3 | 5.2
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Comparison of percentage difference between ezetimibe and placebo; Test type: Superiority or Other; p = 0.365, Fisher Exact

6. Secondary Outcome: Percent Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline
Description: LDL-C levels measured at baseline and after 24 weeks of treatment
Time Frame: Baseline and Week 24
Population: Full Analysis Set (FAS) defined as all enrolled participants who received at least 1 dose of study drug and baseline and follow-up data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 74 | 76
Percent Change | -22.79 [-25.81 to -19.78] | -1.75 [-4.73 to 1.24]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal analysis of covariance; [statistical method as in outcome 1, analysis 1]; Difference in Least-squares Means = -21.05, 95% CI 2-sided [-25.06 to -17.03] — ezetimibe minus placebo

7. Secondary Outcome: Percent Change in Total Cholesterol (TC) From Baseline
Description: TC levels measured at Baseline and after 24 weeks of treatment.
Time Frame: Baseline and Week 24
Population: FAS defined as all enrolled participants who received at least 1 dose of study drug and baseline and follow-up data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 74 | 76
Percent Change | -15.01 [-17.34 to -12.68] | -1.47 [-3.77 to 0.84]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal analysis of covariance; [statistical method as in outcome 1, analysis 1]; Difference in Least-squares Means = -13.54, 95% CI 2-sided [-16.66 to -10.42] — ezetimibe minus placebo

8. Secondary Outcome: Percent Change in Triglycerides From Baseline
Description: Triglycerides levels measured at baseline and after 24 weeks of treatment.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 74 | 76
Percent Change | -7.52 [-14.97 to -0.08] | 3.83 [-3.57 to 11.23]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.025, Longitudinal Analysis of Covariance; [statistical method as in outcome 1, analysis 1]; Difference in Least-squares Means = -11.36, 95% CI 2-sided [-21.27 to -1.44] — ezetimibe minus placebo

9. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline
Description: HDL-C levels measured at baseline and after 24 weeks of treatment.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 74 | 76
Percent Change | 3.86 [0.77 to 6.96] | 1.41 [-1.64 to 4.47]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.246, Longitudinal Analysis of Covariance; [statistical method as in outcome 1, analysis 1]; Difference in Least-squares Means = 2.45, 95% CI 2-sided [-1.71 to 6.61] — ezetimibe minus placebo

10. Secondary Outcome: Percent Change in Non-HDL-cholesterol From Baseline
Description: Non-HDL-C levels measured at baseline and after 24 weeks of treatment.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 74 | 76
Percent Change | -21.32 [-24.05 to -18.59] | -2.25 [-4.95 to 0.45]
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal Analysis of Covariance; [statistical method as in outcome 1, analysis 1]; Difference in Least-squares Means = -19.07, 95% CI 2-sided [-22.71 to -15.43] — ezetimibe minus placebo

ADVERSE EVENTS:
Time Frame: up to 24 weeks for non-serious adverse events (AEs); up to 28 weeks for serious AEs
Description: All Subjects Treated (AST) Population defined as all participants who received at least 1 dose of study drug.
Arm/Group | Ezetimibe | Placebo
Serious Adverse Events (participants affected / at risk) | 2/75 | 5/77
Other Adverse Events (participants affected / at risk) | 17/75 | 25/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe (N=75) | Placebo (N=77)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 1 (2) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe (N=75) | Placebo (N=77)
NASOPHARYNGITIS (Infections and infestations) | 11 (12) | 13 (15)
PHARYNGITIS (Infections and infestations) | 0 (0) | 4 (6)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 (8) | 7 (14)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 7 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.